CLINICAL TRIAL: NCT06424002
Title: The Impact, Feasibility Acceptability and Cost Effectiveness of the RTS,S/AS01 Malaria Vaccine in School Aged Children
Brief Title: The Impact RTS,S/AS01 Vaccine in School Aged Children RTS,S/AS01 Malaria Vaccine in School Aged Children
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Kamuzu University of Health Sciences (Other)
Collaborators: Ministry of Health, Malawi (Other Government); Boston University (Other); Michigan State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P.09/22/3771
Record Dates: First submitted 2023-02-22; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RTS,S/AS01 Vaccine (Experimental): Three doses of the vaccine will be administered, each with one month interval. RTS,S is a subunit vaccine that includes a portion of the circumsporozoite protein (CSP) co-expressed with Hepatitis B surface antigen. The adjuvant is AS01.
  Interventions: Biological: Mosquirixs
- RTS,S/AS01 Vaccine plus artemether-lumefantrine (Experimental): RTS,S/AS01 Vaccine will be provided with a therapeutic dose of artemether-lumefantrine (20 mg of artemether and 120 mg of lumefantrine). Artemether-lumefantrine will be given twice a day for 3 days based on the weight of the child as per treatment guidelines.
  Interventions: Biological: Mosquirixs; Drug: artemether-lumefantrine
- Artemether-lumefantrine only (Experimental): A therapeutic dose of artemether-lumefantrine will be given twice a day for 3 days based on the weight of the child as per treatment guidelines.
  Interventions: Drug: artemether-lumefantrine
- Vitamin A (No Intervention): This is the control group where Vitamin A will be given.

INTERVENTIONS:
Biological: Mosquirixs — RTS,S is a subunit vaccine that includes a portion of the circumsporozoite protein (CSP) co-expressed with Hepatitis B surface antigen. The adjuvant is AS01. Three doses of the vaccine will be administered, each with one month interval.
  Arms: RTS,S/AS01 Vaccine; RTS,S/AS01 Vaccine plus artemether-lumefantrine
Drug: artemether-lumefantrine — A therapeutic dose of artemether-lumefantrine (20 mg of artemether and 120 mg of lumefantrine) will be given twice a day for 3 days based on the weight of the child as per treatment guidelines.
  Arms: Artemether-lumefantrine only; RTS,S/AS01 Vaccine plus artemether-lumefantrine

SUMMARY:
Across sub-Saharan Africa, school-age children bear an under-appreciated burden of malaria. An estimated 200 million school-age children are at risk of malaria and in many areas prevalence of infection exceeds 50%. The high infection rates in this group serves as a source of onward parasite transmission, undermining elimination and control efforts. Furthermore, malaria illness and malaria-induced anemia in this age group lead to school absenteeism, and impaired cognitive function and classroom attention, ultimately resulting in reduced academic achievement. Although universal malaria interventions, such as insecticide treated nets (ITNs) and access to prompt diagnosis and treatment are available to school-age children, this age group is the least likely to benefit from these interventions. Furthermore, efficacy of these approaches may be compromised by increasing anti-malarial drug and insecticide resistance. A malaria vaccine could help to avert the burden of malaria in this age group.

The RTS,S/AS01 malaria vaccine has recently been recommended for vaccination of young children (< 24 months) by the World health organization (WHO) after a Phase 3 trial and an implementation trial showed that the vaccine had moderate but significant efficacy to prevent clinical and severe malaria in young children. Previous randomized trials suggest that the vaccine is safe for older children. However, efficacy of the vaccine has never been assessed in school age children. Kamuzu University of Health Sciences in partnership with the Malawian Ministry of Health seeks to evaluate the efficacy of the newly introduced RTSS/AS01 malaria vaccine in school aged children. The study hypothesizes that vaccination will decrease the morbidity and transmission of malaria, as well as improve school absenteeism and educational outcomes.

DETAILED DESCRIPTION:
This study will be an individual randomized open-label clinical trial to assess the impact, feasibility, acceptability and cost effectiveness of the RTS,S/AS01 vaccine in school-aged children in a malaria endemic environment.

A total of 5400 children aged 6 to 15 years who are attending standards 1-8 in five schools in rural (Machinga) district of Malawi will be randomized to one of the four intervention arms: RTS,S/AS01 vaccine only (RTS,S-only), RTS,S/AS01 vaccine plus an effective antimalarial (artemether-lumefantrine) at the start of the study (RTS,S+AL), artemether-lumefantrine only (AL-only) and a control group that receives only Vitamin A at the start of the study (VIT-A). After obtaining consent from guardians and assent from children older than 13 years of age, participating children will be randomly allocated in a 1:1:1:1 ratio into the intervention arms. Randomization will be stratified by classroom and school. Additionally, two siblings of a subset of 1000 children receiving the vaccine will be enrolled to evaluate the indirect effect of vaccination.

All children will be followed for up to 12 months after vaccination. Clinical malaria will be ascertained through passive case detection (PCD), and attendance and education outcomes will be ascertained through school records. PCD will conducted using the Learner Treatment Kit program platform, a school-based malaria diagnosis and treatment program that the Ministry of Health and Education are currently supporting across the selected schools. Through PCD, the safety of the interventions will also be monitored.

In a subset of 1000 enrolled in the study (250 per intervention arm) and two of their siblings will also be followed in three pre-scheduled visits, the active case detection (ACD) cohort in which the investigators will evaluate outcomes including the direct effect of the vaccine on malaria subclinical infection and the indirect effect of the vaccine. Children will be selected for this cohort randomly, stratifying the samples by school and four age strata (6-7 years, 8-9 years, 10-12 years, 13-15 years). Participants will be invited to visit a health center at baseline, i.e., before the interventions are administered, one month, six months, and 12 months after the end of the primary regimen of RTS,S/AS01. At each of these visits, capillary blood (~500 µl) will be collected through finger pricks for a dry blood spot, from which malaria quantitative polymerase chain reactions (qPCRs) will be performed to detect asexual parasites. In addition, one drop of blood will be used to measure hemoglobin concentrations. The remaining blood will be stored In 500 children enrolled in the ACD cohort and receiving vaccination, 6 mL of venous blood will be collected to evaluate immunological outcomes. These children will be randomly selected among those receiving RTS, S/AS01 (200 RTSS+AL and 200 RTSS-only) in four schools (50 X 2 intervention groups in each school), and the 4 age strata (~ 12 per age strata in each school and intervention group).

Feasibility, acceptability and cost data will be collected through interviews with all study stakeholders: learners, parents, teachers, community leaders, and district and national policy makers.

ELIGIBILITY:
Inclusion criteria:

* Pupils aged approximately 6 years to 15 years and enrolled in Standard 1 - 8 in the participating schools
* Planning to remain in the study area for 1 year
* Parental/guardian consent for child's participation and child assent if the child is 13 years of age or older

Exclusion criteria:

* Pregnancy, defined based on menstrual history. Pupils who had their last menstrual period more than 6 weeks before enrollment will be excluded. This threshold was chosen considering that menstrual cycles are irregular in this age group
* Viral infections resulting in fever, chills, new loss of taste/smell and sore throat
* Known allergy or history of adverse reaction to antimalarial treatment or vaccines
* Chronic use of anti-malarial medication, azithromycin, or cotrimoxazole
* Enrollment in any other study
* Evidence of heart disease, HIV, or epilepsy
* Severe disability

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5400 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled school children with clinical malaria incident events throughout the study period (PCD). | During 18 months of follow up, when the child presents with symptoms of malaria within 48 hours at the leaner treatment kit (LTK) program which is run by teachers
  Based on symptoms of malaria plus a positive malaria rapid diagnostic test. A bood slide will also be collected for future assessment for malaria parasites
Proportion of enrolled school children that are daily absent from class throughout the study period (using electronic classroom registers) | During 18 months of follow up, a daily register will be administered to record school attendance
  This will be based on electronic classroom registers

SECONDARY OUTCOMES:
Proportion of enrolled school children who pass their examinations at the end of the year and proceed to the next class (Pupil's passing fraction based on classroom records) | During 18 months of follow up, classroom records will record children passing end of year examinations
  Pass rate based on classroom records
Proportion of enrolled school children with clinical malaria incident events throughout the study period (ACD) | During 18 months of follow up, clinical malaria will be assessed during sick visits (PCD) and during active case detection
  Based on symptoms of malaria plus a positive malaria rapid diagnostic test. A bood slide will also be collected for future assessment for malaria parasites
Proportion of enrolled school children with P. falciparum infections during the study period (ACD). | During 18 months of follow up, malaria infection will be assessed during the ACD visits
  Based dried blood spot (DBS) samples from index child
Proportion of children with low levels of hemoglobin levels (hb<11g/dl) during the study period (ACD). | At baseline, midline, endline and during ACD visits, hemoglobin levels will be measured during the 18 months follow up period
  As measured by hemocue machines
Proportion of siblings of enrolled children with P. falciparum infections at the beginning and end of the study period (indirect or "spill over" effect) (ACD) | During 18 months of follow up, malaria infection will be assessed during the ACD visits
  Based DBS samples from siblings of index child
Levels of antibodies against N-4-azido-2-nitrophenylpyridoxyl-5-phosphate (NANP) and CSP | At endline and during ACD visits, levels of antibodies will be measured during 18 months of follow up
  Magnitude of immunoglobulin G (IgG) against NANP. 2. Geometric mean of magnitude of antibodies against the two antigens, as well as avidity, and fractional catabolic rate (FcR) binding activity over time.

CONTACTS AND LOCATIONS:
Overall Officials: Don P Mathanga, PhD, Principal Investigator — Kamuzu University of Health Sciences

IPD SHARING:
Plan to Share IPD: Yes
Under this proposal, Investigators will de-identify all the data intended for broader use, and all variables that could be used to deductively disclose the identity of individual subjects. Examples of data that will be removed include names, dates of birth, medical record numbers, telephone numbers, and locations of homes.
  All data will be sent to the approved Malawi government data repository center for safe keeping and will also be made available through NIH-supported portals for wide dissemination and access. Any data shared will be subject to Malawi government conditions of use governing access to the public release of data, including restrictions against attempting to identify study participants, destruction of data after analyses are completed, reporting responsibilities, restrictions on redistribution of data to third parties, and proper acknowledgement of data source.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study
Access Criteria: Access will be based on requests and review of the request. As per NIH policy, data will be shared through approved links.